CLINICAL TRIAL: NCT03654209
Title: Prospective Randomized Controlled Trial Describing the Recurrence Rate of Adenomas in Sessile or Flat Colonic Lesions 15mm or Larger Receiving Post-resection Site Treatment With Snare Tip Soft Coagulation or Argon Plasma Coagulation
Brief Title: Post-resection Treatment of Large Colon Polyps
Acronym: SAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Erbe USA Incorporated (Other)
Responsible Party: Principal Investigator, Douglas K. Rex, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1805411306; NCT04063280 (obsolete NCT alias)
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Recurrence
Keywords: Argon Plasma Coagulation; Snare Tip Soft Coagulation; Recurrence rates
MeSH Terms: conditions — Recurrence | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to Argon Plasma Coagulation vs Snare Tip Soft Coagulation vs no treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Argon Plasma Coagulation (Experimental): Following polyp removal using standard of care methods, Argon Plasma Coagulation (APC) will be applied to the perimeter of the resection site before any clips are added.
  Interventions: Device: Argon Plasma Coagulation
- Snare Tip Soft Coagulation (Experimental): Following polyp removal using standard of care methods, Snare Tip Soft Coagulation (STSC) will be applied to the perimeter of the resection site before any clips are added.
  Interventions: Device: Snare Tip Soft Coagulation
- No treatment (No Intervention): Following polyp removal using standard of care methods, neither APC nor STSC will be applied to the perimeter of the resection site. Clips may be added at the discretion of the PI.

INTERVENTIONS:
Device: Argon Plasma Coagulation — APC will be applied to the perimeter of the resection site
  Arms: Argon Plasma Coagulation
Device: Snare Tip Soft Coagulation — STSC will be applied to the perimeter of the resection site
  Arms: Snare Tip Soft Coagulation

SUMMARY:
Patients who have provided informed consented and are scheduled to undergo endoscopic mucosal resection (EMR) of lesions 15mm and larger will be randomized to STSC (80 W, Effect 5) vs APC (preferred settings) vs No Treatment of the perimeter of the EMR site.

DETAILED DESCRIPTION:
Data regarding polyp morphology, location & shape will be recorded in addition to procedure and treatment length. Injection fluid use and clipping will also be recorded in addition to any procedural complications.

All randomized subjects will receive a 30-day post procedure follow-up phone call and be scheduled, as per the standard of care, to receive a standard follow-up colonoscopy procedure after the initial procedure. The investigators will measure the rate of recurrence by endoscopic visualization of the EMR site at the first follow-up using endoscopic magnification and electronic chromoendoscopy, as well as systematic biopsy of the scars.

ELIGIBILITY:
Inclusion Criteria:

* 25 years and older
* Ability to provide informed consent
* Undergoing colonoscopy for screening, surveillance, diagnostic reasons, or removal of a lesion

Exclusion Criteria:

* Pedunculated lesions
* Inflammatory bowel disease
* Inability to provide informed consent
* Lesions less than 15mm in largest dimension

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K. Rex, MD, Principal Investigator — Indiana University
Locations (10):
- United States (10):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Orlando, Orlando, Florida
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Spring Mill Medical Center, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
De-identified data can be shared in the future upon request.

REFERENCES:
- [Background] Zhan T, Hielscher T, Hahn F, Hauf C, Betge J, Ebert MP, Belle S. Risk Factors for Local Recurrence of Large, Flat Colorectal Polyps after Endoscopic Mucosal Resection. Digestion. 2016;93(4):311-7. doi: 10.1159/000446364. Epub 2016 Jun 7. PMID 27271329
- [Background] Brooker JC, Saunders BP, Shah SG, Thapar CJ, Suzuki N, Williams CB. Treatment with argon plasma coagulation reduces recurrence after piecemeal resection of large sessile colonic polyps: a randomized trial and recommendations. Gastrointest Endosc. 2002 Mar;55(3):371-5. doi: 10.1067/mge.2002.121597. PMID 11868011
- [Background] Tate DJ, Bahin FF, Desomer L, Sidhu M, Gupta V, Bourke MJ. Cold-forceps avulsion with adjuvant snare-tip soft coagulation (CAST) is an effective and safe strategy for the management of non-lifting large laterally spreading colonic lesions. Endoscopy. 2018 Jan;50(1):52-62. doi: 10.1055/s-0043-119215. Epub 2017 Oct 11. PMID 29020690
- [Derived] Rex DK, Haber GB, Khashab M, Rastogi A, Hasan MK, DiMaio CJ, Kumta NA, Nagula S, Gordon S, Al-Kawas F, Waye JD, Razjouyan H, Dye CE, Moyer MT, Shultz J, Lahr RE, Yuen PYS, Dixon R, Boyd L, Pohl H. Snare Tip Soft Coagulation vs Argon Plasma Coagulation vs No Margin Treatment After Large Nonpedunculated Colorectal Polyp Resection: a Randomized Trial. Clin Gastroenterol Hepatol. 2024 Mar;22(3):552-561.e4. doi: 10.1016/j.cgh.2023.09.041. Epub 2023 Oct 21. PMID 37871841

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Argon Plasma Coagulation | Snare Tip Soft Coagulation | No Treatment
Started | 126 | 126 | 132
Completed | 103 | 100 | 105
Not Completed | 23 | 26 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Argon Plasma Coagulation | Snare Tip Soft Coagulation | No Treatment | Total
Number analyzed (Participants) | 126 | 126 | 132 | 384
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (9.7) | 66.0 (9.8) | 65.5 (10.1) | 65.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 55 | 49 | 162
  Male | 68 | 71 | 83 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 2 | 10
  Not Hispanic or Latino | 120 | 124 | 127 | 371
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 4 | 11 | 23
  White | 114 | 117 | 112 | 343
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 126 | 126 | 132 | 384
Boston Bowel Prep Score [Median (Inter-Quartile Range); unit: scores on a scale] — Boston Bowel Preparation Score for patients. The total score for the Boston Bowel Preparation Scale ranges from 0 to 9, with higher score indicating a better bowel preparation quality.
  scores on a scale | 9 [7 to 9] | 9 [8 to 9] | 9 [8 to 9] | 9 [8 to 9]
Follow-up Colonoscopy Interval [Median (Inter-Quartile Range); unit: Months] | 6.4 [6.0 to 8.0] | 6.4 [6.0 to 10.7] | 6.3 [6.0 to 8.3] | 6.4 [6.0 to 8.7]
Site [Count of Participants; unit: Participants]
  AdventHealth Orlando | 18 | 16 | 19 | 53
  Dartmouth-Hitchcock Medical Center | 3 | 4 | 2 | 9
  Indiana University | 41 | 42 | 43 | 126
  Johns Hopkins Hospital | 14 | 14 | 15 | 43
  Mount Sinai Hospital | 17 | 17 | 16 | 50
  NYU Langone Medical Center | 20 | 21 | 23 | 64
  Penn State Health Milton S. Hershey Medical Center | 1 | 1 | 2 | 4
  Sibley Memorial Hospital | 2 | 2 | 2 | 6
  The University of Kansas Medical Center | 10 | 9 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Recurrence
Description: The recurrence rate of adenomas at the site of any qualifying, previously resected lesions will be measured at the first follow-up colonoscopy
Time Frame: 1 day
Population: There were 103 patients that completed follow-up colonoscopy in the APC arm of the study. Since some patients had more than one eligible polyp for the study, there ended up being 108 lesions assessed for recurrence in the APC arm. For the same reason, there are 100 patients but 108 polyps in the STSC group and 105 patients but 112 polyps in the No Treatment group.
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Argon Plasma Coagulation | Snare Tip Soft Coagulation | No Treatment
Number analyzed (Participants) | 103 | 100 | 105
Number analyzed (Polyps) | 108 | 108 | 112
Polyps | 10 | 5 | 24

2. Primary Outcome: Types of Recurrences
Description: Description of whether recurrence was visible during the follow-up procedure and confirmed by pathology, visible during the follow-up procedure but not confirmed by pathology, or not visible during the follow-up procedure but confirmed by pathology of biopsies taken.
Time Frame: 1 day
Population: There were 103 patients that completed follow-up colonoscopy in the APC arm of the study. Since some patients had more than one eligible polyp for the study, there ended up being 108 lesions assessed to check for recurrence in the APC arm. For the same reason, there are 100 patients but 108 polyps in the STSC group and 105 patients but 112 polyps in the No Treatment group.
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Argon Plasma Coagulation | Snare Tip Soft Coagulation | No Treatment
Number analyzed (Participants) | 103 | 100 | 105
Number analyzed (Polyps) | 108 | 108 | 112
Polyps
  Visible recurrence - Pathology verified | 8 | 5 | 15
  Not visible recurrence - Pathology positive | 2 | 0 | 8
  Visible recurrence - No pathology verification | 0 | 0 | 1

3. Secondary Outcome: Time
Description: The time it takes to apply each respective treatment (APC or STSC) on the day of procedure
Time Frame: 1 day
Population: There were 126 patients in the APC arm of the study. Since some patients had more than one eligible polyp for the study, there ended up being 134 lesions included in the APC arm. For the same reason, there are 126 patients but 140 polyps in the STSC group and 132 patients but 140 polyps in the No Treatment group.
Measure: Median (Inter-Quartile Range); unit: Minutes
Units Other Than Participants: Polyps
Arm/Group | Argon Plasma Coagulation | Snare Tip Soft Coagulation | No Treatment
Number analyzed (Participants) | 126 | 126 | 132
Number analyzed (Polyps) | 134 | 140 | 140
Minutes | 4.08 [2.75 to 6.40] | 3.35 [1.97 to 6.00] | NA [NA to NA] — The No Treatment arm did not receive margin treatment, so the time to apply margin treatment is not applicable for this group.

4. Secondary Outcome: Complications
Description: To look at the number of complications for each randomization arm as assessed through a 30 day follow-up period
Time Frame: 1 day
Population: Number of patients that completed the follow-up to collect adverse event information.
Measure: Number; unit: Adverse Events
Arm/Group | Argon Plasma Coagulation | Snare Tip Soft Coagulation | No Treatment
Number analyzed (Participants) | 116 | 122 | 123
Adverse Events
  Delayed Bleeding | 3 | 4 | 6
  Perforation | 0 | 0 | 0
  Post Polypectomy Syndrome | 0 | 1 | 1
  Myocardial Infarction | 1 | 0 | 0
  Hospitalization | 3 | 5 | 6

ADVERSE EVENTS:
Time Frame: 1 month
Description: Patients were called approximately 30 days after their colonoscopy procedure.
Arm/Group | Argon Plasma Coagulation | Snare Tip Soft Coagulation | No Treatment
All-Cause Mortality (participants affected / at risk) | 1/126 | 0/126 | 0/132
Serious Adverse Events (participants affected / at risk) | 7/126 | 10/126 | 13/132
Other Adverse Events (participants affected / at risk) | 27/126 | 30/126 | 24/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Argon Plasma Coagulation (N=126) | Snare Tip Soft Coagulation (N=126) | No Treatment (N=132)
Delayed Bleeding (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 6 (6)
Post Polypectomy Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Argon Plasma Coagulation (N=126) | Snare Tip Soft Coagulation (N=126) | No Treatment (N=132)
Intraprocedural bleed during index polyp removal (Injury, poisoning and procedural complications) | 13 (15) | 14 (14) | 16 (16)
Type 3 Muscle Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Pain (Injury, poisoning and procedural complications) | 4 (4) | 12 (12) | 3 (3)
Delayed Bleeding (Injury, poisoning and procedural complications) | 8 (8) | 8 (8) | 2 (2)
Bowel Movement Irregularity (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Anesthesia Reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombosed AV fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Blood clots (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Paracentesis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nose bleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post-Polypectomy Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Imbalance in patient recruitment among sites. We included polyps resected en bloc & 15-19mm polyps. Whether margin treatment is beneficial after en bloc resection or removal of 15-19 mm polyps is unknown.

Endoscopists couldn't be blinded to randomized treatment. Dropout rate was higher than expected, so planned power was slightly reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/09/NCT03654209/Prot_SAP_000.pdf